CLINICAL TRIAL: NCT05991986
Title: Production of Patient Autologous Induced Pluripotent Stem Cell-derived Retinal Cells for Age-related Macular Degeneration
Brief Title: Preparation of Patient Autologous Induced Pluripotent Stem Cell-derived Retinal Cells for AMD
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiufeng Zhong, Prof, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2023KYPJ224
Record Dates: First submitted 2023-07-26; First posted 2023-08-15 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — somatic cells isolated from urine, peripheral blood, skin biopsies, conjunctiva biopsies, etc.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: somatic cell collection — One or more types of somatic cells will be collected from every participant by collecting approximately 100~500 ml of midstream urine, 20~30 ml of peripheral blood, skin biopsies (3mm), conjunctiva biopsies (5mm×5mm), etc.

SUMMARY:
This project intends to collect participant somatic cells to prepare autologous induced pluripotent stem cell-derived retinal cells for future cell therapy of age-related macular degeneration patient.

DETAILED DESCRIPTION:
One or more types of somatic cells will be collected from every participant by collecting approximately 100~500 ml of midstream urine, 20~30 ml of peripheral blood, skin biopsies (3mm), conjunctiva biopsies (5mm×5mm), etc. Then, these somatic cells will be used to prepare patient autologous induced pluripotent stem cell-derived retinal cells for the cell therapy of age-related macular degeneration patient.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 55-80 years;
2. Clinical diagnosis is consistent with the definition of advanced age-related macular degeneration;
3. The BCVA of the target eye will be lower than 20/200;
4. -8.00 D < refraction < +8.00 D, 21 mm < anteroposterior axis≤ 28 mm;
5. Voluntary as test subjects, informed consent, regular follow-up on time;
6. Voluntary as test subjects to join the associated clinical research on autologous iPSC-derived retinal cell therapy for AMD (ethical approval and informed consent documents will be applied and signed separately);

Exclusion Criteria:

1. Macular atrophy caused by other diseases in addition to AMD;
2. Malignant tumor and history of malignancy;
3. Any immune deficiency;
4. Lens opacities (affecting the central vision), glaucoma, uveitis, retinal detachment, inherited retinal dystrophy, optic neuropathy, and other ocular histories;
5. Other intraocular surgery histories besides cataract surgery;
6. Severe heart failure or the left ventricular ejection fraction <35% in the previous 6 months;
7. Dialysis or eGFR <20ml/min/1.73m2;
8. Urine protein/urine creatinine ratio ≥1g/g;
9. Creatinine or albumin/urine creatinine ratio ≥600mg/g;
10. Chronic liver disease with ALT three times over the upper limit of normal value;
11. Combined with severe systemic diseases, such as heart failure, liver disease, COPD, etc.
12. Combined with severe infectious diseases, such as HIV, HBV, HCV, syphilis, etc.
13. HCV-RNA positive, HBV-DNA >103 IU/ml, or TB, etc., during the infectious period;
14. Use anticoagulant, or the platelet function is still not restored to normal after stopping antiplatelet drugs for 10 days;
15. Abnormal blood coagulation function or other laboratory tests;
16. Use glucocorticoids, immunosuppressive drugs, or antipsychotic drugs in the previous 3 months;
17. Use antipsychotic drugs in the previous 3 months, such as antidepressants drugs, antimanic drugs, etc.
18. Allergy to tacrolimus or other macrolides;
19. A history of addiction to alcoholism or prohibited drugs;
20. Be participating in other intervention clinical trials or receiving other study medications;
21. Informed refusal；
22. Some other situations which might increase the risks of the subjects or interfere with clinical trials, such as mental disorders, cognitive dysfunction, etc.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMD patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
somatic cell collection | 2023.8.1~2026.7.31
  somatic cell collection

CONTACTS AND LOCATIONS:
Overall Officials: Xiufeng Zhong, Doctor, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University